CLINICAL TRIAL: NCT03493009
Title: Optimizing the Preparation Regime Prior to Colonoscopy Procedure With Pure-Vu System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties to sign a contract with the hospital, due to logistic changes in the hospital.
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CL00042
Record Dates: First submitted 2017-12-27; First posted 2018-04-10 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2017-12

CONDITIONS: Gastrointestinal Diseases; Colorectal Cancer
MeSH Terms: conditions — Gastrointestinal Diseases; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization in blocks will be applied for each site to allocate patients to one of two different bowel preparation regimens (Prep A- split doae of 10mg of Magnesium citrate versus Prep B- split doae of 15mg of Magnesium citrate). The study will utilize randomization in blocks using the standard envelope procedure, which will be applied in order to allocate patients into two arms:
  * Group 1 - Will go through the Prep A procedure
  * Group 2 - Will go through the Prep B procedure The site randomization plan will be provided to the study coordinator prior the study start.
Masking Description: No blinding is applicable in this study .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10mg Magnesium citrate (Experimental): subjects will be required to follow a specific bowel preparation instruction consisting of dietary restrictions (no dried fruit, seeds or nuts) starting 5 days prior to the colonoscopy, an low residue diet at the day before the procedure, followed by a split dose of 10 mg of Magnesium citrate, followed by colonoscopy procedure with Pure-Vu System
  Interventions: Device: Pure-Vu System
- 15mg Magnesium citrate (Experimental): subjects will be required to follow a specific bowel preparation instruction consisting of dietary restrictions (no dried fruit, seeds or nuts) starting 5 days prior to the colonoscopy, an low residue diet at the day before the procedure, followed by a split dose of 15 mg of Magnesium citrate, followed by colonoscopy procedure with Pure-Vu System
  Interventions: Device: Pure-Vu System

INTERVENTIONS:
Device: Pure-Vu System — The Pure-Vu System is Food and Drug Administration (FDA) approved device since September 22, 2016, intended to connect to standard colonoscopes to help facilitate intra-procedural cleaning of a poorly prepared colon by irrigating or cleaning the colon and evacuating the irrigation fluid (water), feces and other bodily fluids and matter, e.g. blood.

SUMMARY:
The primary objective of this multicenter, prospective, randomized study is to evaluate the performance of Pure-Vu System in cleansing patients' colon who are indicated for a colonoscopy procedure using one of two different reduce bowel preparation regimes.in addition, the cecum intubation rate, time to cecum, total procedure time, and adverse event will be evaluated.

DETAILED DESCRIPTION:
This multicenter, prospective, randomized study will include up to 100 patients (30 patients per site and 15 patients per study arm), aimed at evaluating the performance of Pure-Vu System in cleansing patients' colon who are indicated for colonoscopy procedure using one of two different preparation regimes as detailed below.

Subjects will be enrolled at up to 10 clinical sites in the United States. Subjects who meet the eligibility criteria will be randomly allocated to a given study arm and will be required to follow a specific bowel preparation instruction along with a specific prep agent (Bowel preparation instructions for morning and afternoon procedures are provided in appendix B1 and B2, respectively), as per study arm allocation, starting 5 days prior to the colonoscopy with Pure-Vu. Patients will be asked to record and provide their diet and bowel movements in the provided diary log at time of their scheduled colonoscopy (Diary log is provided in appendix D).

In addition patient will be ask to complete a satisfaction questionnaire include feedback on the procedure and on specific aspects related to the preparation regime.

Following the procedure a telephone follow-up will be conducted at 48 hours (± 48 hours) post Pure-Vu procedure to assess patient well-being and capture any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled for colonoscopy procedure
2. Subjects in the age range of 22-75 years inclusive
3. Subject is willing and able to participate in the study procedures and to understand and sign the informed consent.

Exclusion Criteria:

1. Patients with active Inflammatory Bowel Disease
2. Patients with known diverticulitis disease or with prior incomplete colonoscopy due to diverticular disease
3. Patients with known bowel obstruction
4. Patient with chronic constipation
5. History of prior surgery to colon and/or rectum
6. ASA (Physical status classification system) ≥ III
7. Renal insufficiency (Creatinine ≥ 1.5mg /dL) (based on medical history)
8. Abnormal Liver enzymes (ALT/AST ≥ 2 times upper limits of normal) (based on medical history)
9. Patients taking anticoagulants drugs (excluding aspirin) or dual antiplatelet therapy
10. Patients with known coagulation disorder (INR >1.5).
11. Pregnancy (as stated by patient) or breast feeding
12. Patients with altered mental status/inability to provide informed consent

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
rate of adequate cleansing level | up to 2 hours
  The rate of adequate cleansing level in each colon segment before and after use of Pure-Vu will be evaluated per study arm using the Boston Bowel Preparation Scale (BBPS). Segment score of 0-3 given to each of the 3 segments of the colon (Left side, Transverse and right side).
  BBPS* scores will be rated by the colonoscopies, on the basis of three segment scores summed for maximum score of 9, where:
  * 0 = unprepared
  * 9 = completely clean (in completed to Cecum procedures) An adequate cleansing procedure will be considered when all the colon segments will be graded as 2 or above.

IPD SHARING:
Plan to Share IPD: Undecided
no plan to share the individual participated date with other researchers at this point.

DOCUMENTS (1):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT03493009/Prot_000.pdf